CLINICAL TRIAL: NCT00291447
Title: A Phase 1 Single Dose Escalation Trial of ch806 in Patients With Advanced Tumours Expressing the 806 Antigen
Brief Title: 111In-ch806 in Patients With Advanced Tumours Expressing the 806 Antigen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LUD2004-001
Record Dates: First submitted 2006-02-10; First posted 2006-02-14 (Estimated); Results first posted 2021-06-08 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — monoclonal antibody 806

STUDY DESIGN:
Intervention Model Description: Open label, single dose escalation Phase I trial of ch806 in patients with advanced tumors expressing the 806 antigen.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Patients received a single infusion of 5 mg/m2 111In-ch806 on Day 0 and followed for 30 days post infusion.
  Interventions: Biological: ch806
- Cohort 2 (Experimental): Patients received a single infusion of 10 mg/m2 111In-ch806 on Day 0 and followed for 30 days post infusion.
  Interventions: Biological: ch806
- Cohort 3 (Experimental): Patients received a single infusion of 20 mg/m2 111In-ch806 on Day 0 and followed for 30 days post infusion.
  Interventions: Biological: ch806
- Cohort 4 (Experimental): Patients received a single infusion of 40 mg/m2 111In-ch806 on Day 0 and followed for 30 days post infusion.
  Interventions: Biological: ch806

INTERVENTIONS:
Biological: ch806 — ch806 is a chimeric (part human, part mouse) antibody which recognizes and attaches to a protein called the 806 antigen (a type of EGFR), which is found on the surface of some cancer cells.

SUMMARY:
The purpose of this clinical trial is to describe the toxicity, biodistribution, pharmacokinetics and tumour uptake of a single infusion of ch806 (tagged with a trace amount of radioactive 111-Indium: 111In-ch806) in patients with advanced tumours expressing the 806 antigen.

DETAILED DESCRIPTION:
This clinical research study explores the activity of the new experimental antibody ch806 in humans for the first time.

Cancers arising from an organ can be cured in some cases with various combinations of surgery, chemotherapy and radiotherapy. However, once some cancers spread to other organs, treatment with commonly used methods is unlikely to cure the cancer and so treatment is then designed to control the growth of the cancer, and the problems it is causing. One newer treatment approach involves targeting a marker (antigen) called the epidermal growth factor receptor (EGFR), which is found on the tumour cell's surface, with a specially constructed monoclonal antibody (mAB) called "ch806".

Antibodies are proteins that are found in the blood. Antibodies normally protect us from foreign invaders, such as bacteria or viruses. They help destroy these foreign substances by binding to them and activating white blood cells or blood proteins, resulting in their destruction. Tumour cells also have antigens which can be targeted by antibodies. A receptor expressed in high amounts (over-expressed) on various cancer cells, called the epidermal growth factor (EGFR), has been identified, studied and targeted with a variety of antibodies.

One of these antibodies, monoclonal antibody 806 (mAb806), was originally made from mouse protein. Because mAb806 is a mouse antibody, if it were given to humans the body would see it as a foreign protein and would be likely to react to it with an unwanted immune response. To overcome this, the structure of the original mouse antibody called mAb 806 was changed to appear more "human-like" and the chimeric antibody (part mouse part human) called ch806 was produced.

The study is open to patients whose tumour is shown to express the 806 antigen by a special test. Further tests are required to determine eligibility for the study. These tests determine general health and include: physical examination; blood samples for routine tests; routine tests to determine the extent of tumour prior to starting treatment with 111In-ch806 (eg. X-ray, CT scan, etc.).

On study, 111In-ch806 is given by infusion into a vein over one hour. Blood samples to determine the amount of drug in the blood (pharmacokinetics), are taken a number of times on the day of the 111In-ch806 infusion; about every 2nd day for the first week; then 2 weeks, 3 weeks and 4 weeks after the infusion. Blood tests are also used to monitor general health and to see if the immune system recognizes the infused antibody by making another antibody against it. Such a response is called "anti-ch806 antibody" or "HACA". Gamma camera scans to see where 111In-ch806 goes in the body are done right after the first infusion, and 4 more times over the next seven days. The scan takes about one hour each time. Visits for weekly follow up examinations and blood tests until 30 days after the infusion are combined with further gamma camera scans. Tumour is reassessed 30 days after the infusion using the same type of scans as at study entry.

Further treatment with a course of 111In-ch806 is not available at this time, as this study is to test the safety of a single infusion only.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced or metastatic tumours which are positive for 806 antigen expression based on chromogenic in situ hybridization (CISH) or immuno-histochemistry (IHC) of archived tumour samples.
* Histologically or cytologically proven malignancy.
* Measurable disease on CT scan with at least one lesion >/= 2 cm diameter (to allow adequate imaging).
* Age greater than or equal to 18 years.
* Karnofsky performance scale >/= 70.
* Within the last 2 weeks vital laboratory parameters should be within normal range, except for the following laboratory parameters, which should be within the ranges specified: Neutrophil count >/= 1.5 x 10^9/L; Platelet count >/= 150 x 10^9/L; Serum bilirubin < 34 micromol/L; Creatinine clearance > 50ml/min
* Able and willing to give valid written informed consent.

Exclusion Criteria:

* Untreated active metastatic disease to the central nervous system (new or enlarging lesions on CT or MRI), or within 3 months of treatment (i.e. surgery or radiotherapy) for brain metastases. Primary central nervous system tumour (e.g. Glioblastoma Multiforme) is not an exclusion criterion.
* Other serious illnesses, e.g., serious infections requiring antibiotics, bleeding disorders.
* Chemotherapy, radiation therapy, or immunotherapy within 4 weeks before study entry (6 weeks for nitrosoureas).
* Clinically significant cardiac disease (New York Heart Association Class III/IV).
* Other malignancy within 3 years prior to entry into the study, except for treated non-melanoma skin cancer and cervical carcinoma in situ.
* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
* Lack of availability for immunological and clinical follow-up assessments.
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.
* Pregnancy or breastfeeding.
* Women of childbearing potential: Refusal or inability to use effective means of contraception.
* Concomitant treatment with systemic corticosteroids except for patients with Glioblastoma. (Topical or inhalational corticosteroids are permitted.)
* Prior administration of monoclonal antibody or antibody fragment, and positive human anti-chimeric antibody (HACA) titre.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-05 (Actual); Primary Completion 2006-02-16 (Actual); Study Completion 2006-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof Andrew M Scott, MBBS MD DDU, Principal Investigator — Ludwig Institute for Cancer Research
Locations (1):
- Ludwig Institute Tumor Targeting Program, Austin Health, Heidelberg, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 1 | 4
  >=65 years | 1 | 1 | 1 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 1
  Male | 2 | 1 | 2 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 2 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 1 | 2 | 7
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Australia | 2 | 2 | 2 | 2 | 8
Karnofsky performance status [Count of Participants; unit: Participants] — 80-100% Able to carry on normal activity and to work; no special care needed; 50 -70% Unable to work; able to live at home and care for most personal needs; varying amount of assistance needed; 10-40% Unable to care for self; requires equivalent of institutional or hospital care; disease may be progressing rapidly.
  Participants
    80-100% | 2 | 2 | 2 | 2 | 8
    50-70% | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events
Description: All AEs occurring during the study were documented on the respective case report form (CRF) pages. Events, which occurred after signed informed consent, but before first administration of study drug, were documented on the Pre-existing Signs and Symptom page. Thereafter, they were documented on the Adverse Event page.
  Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0.
  Documentation of AEs includes: date and time of onset and resolution, severity, frequency, seriousness, related interventions and outcome.
  Dose limiting toxicity (DLT) was defined as any Grade 2 or greater allergic reaction related to 111In-ch806 antibody protein, and any Grade 4 haematological or Grade 3 or greater non-haematological toxicity except for skin rash, occurring within 30 days of the 111In-ch806 infusion.
Time Frame: 30 days
Population: All patients
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 2 | 2 | 2 | 2
Participants
  Number of patients reporting at least 1 adverse event | 2 | 2 | 2 | 2
  Dose limiting toxicities (DLT) | 0 | 0 | 0 | 0

2. Secondary Outcome: Biodistribution of 111In-ch806 Using Whole Body Clearance Methodology or Biological Halftime (T1/2-biol) Following the First Infusion.
Description: Gamma camera images were acquired on Day 0 (1-4 hours after 111In-ch806 infusion), and on Day 1, Day 2 or 3, Day 4 or 5, and Day 6 or 7 post 111In-ch806 infusion.
  Image analysis was performed by defining regions of interest (ROIs) around the kidneys, liver, spleen and lungs and whole body.
  T1/2-biol was calculated from the whole body anterior and posterior planar images.
  A ROI was calculated to encompass the whole body via a morphological dilation and erosion of a binarized planar image, at a user-defined threshold taken as a percentage (0.9 - 1.5%) of maximum pixel value of the planar image. From each ROI at each time point, the mean counts per pixel per minute was normalised to imaging time point Day 0. From this time-activity curve (TAC), an exponential clearance expression was fitted to obtain effective halftime. This was then corrected for the physical half-life of 111In (67.45 hours) to account for physical decay to obtain the biological halftime.
Time Frame: Day 0 (1-4 hours after 111In-ch806 infusion), and on Day 1, Day 2 or 3, Day 4 or 5, and Day 6 or 7 post 111In-ch806 infusion.
Population: All patients
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 2 | 2 | 2 | 2
hours | 1258 (381) | 931 (649) | 915 (207) | 689 (255)

3. Secondary Outcome: Mean Normal Organ Dosimetry of 111In-ch806 Using Normal Organ Absorbed Dose (mGy/MBq) Following the First Infusion.
Description: Gamma camera images were acquired on Day 0 (1-4 hours after 111In-ch806 infusion), and on Day 1, Day 2 or 3, Day 4 or 5, and Day 6 or 7 following 111In-ch806 infusion.
  Dosimetry analysis was performed for kidney, liver, spleen and lung. Organ radioactivity was estimated from the geometric mean (GM) of anterior and posterior sample region of interest (ROI) counts. Three regions were defined for the organs, a whole organ ROI, a sample organ ROI, and a background ROI.
  Average counts within sample ROIs (counts/pixel) were multiplied by the area of the organ (pixels), determined from the whole organ ROI at the time point. For paired organs,a single organ area was measured and then multiplied by two to find total area. The counts for each organ were corrected for background. A time-activity curve (TAC) was generated and fitted with a single component exponential clearance expression. The number of disintegrations, or cumulated activity, was calculated for each organ.
Time Frame: Day 0 (1-4 hours after 111In-ch806 infusion), and on Day 1, Day 2 or 3, Day 4 or 5, and Day 6 or 7 following 111In-ch806 infusion.
Population: All patients
Measure: Mean (Standard Deviation); unit: mGy/MBq
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 2 | 2 | 2 | 2
mGy/MBq
  Kidney | 0.370 (0.026) | 0.365 (0.068) | 0.359 (0.002) | 0.3428 (0.033)
  Liver | 0.504 (0.016) | 0.652 (0.088) | 0.501 (0.053) | 0.475 (0.064)
  Lungs | 0.152 (0.036) | 0.169 (0.061) | 0.163 (0.001) | 0.156 (0.014)
  Spleen: number analyzed (Participants) | 1 | 2 | 2 | 2
  Spleen | 0.194 (NA) — Patient 001 had splenectomy: therefore, only 1 subject included. | 0.313 (0.035) | 0.450 (0.189) | 0.399 (0.035)

4. Secondary Outcome: Number of Patients With Tumour Uptake of 111In-ch806 Based on Qualitative Assessment of Biodistribution Images and Dosimetry Following the First Infusion.
Description: Whole body gamma camera imaging with anterior and posterior whole body scans using conjugate view methodology were performed for assessment of biodistribution and tumour uptake on Day 0 (1-4 hours after 111In-ch806 infusion), Day 1, Day 2 or 3, Day 4 or 5, and Day 6 or 7 following 111In-ch806 infusion. Target lesions (>2cm) were used to measure uptake of 111In-ch806.
Time Frame: Day 0 (1-4 hours after 111In-ch806 infusion), Day 1, Day 2 or 3, Day 4 or 5, and Day 6 or 7 following 111In-ch806 infusion.
Population: All patients
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 2 | 2 | 2 | 2
Participants | 2 | 2 | 2 | 2

5. Secondary Outcome: Mean Half-life as Measured by Half-life of Initial Phase of Disposition (T½α) and Terminal Phase of Distribution (T½β) of 111In-ch806 Following the First Infusion .
Description: The pharmacokinetics of 111In-ch806 were calculated based on gamma counting of serum samples. Serum samples for pharmacokinetics were collected on Day 0 - pre 111In-ch806 infusion; then at 5 minutes, 60 minutes, 2 hours and 4 hours post 111In-ch806 infusion, Day 1, Day 2 or 3, Day 4 or 5, Day 6 or 7, Day 14 (± 2 days) and Day 21 (± 2 days) and Day 30 (± 2 days) post infusion.
Time Frame: Day 0 - pre 111In-ch806 infusion; then at 5 minutes, 60 minutes, 2 hours and 4 hours post 111In-ch806 infusion, Day 1, Day 2 or 3, Day 4 or 5, Day 6 or 7, Day 14 (± 2 days) and Day 21 (± 2 days) and Day 30 (± 2 days) post infusion.
Population: All patients
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Cohort 2: Patients received a single infusion of 10 mg/m2 111In-ch806 on Day 0 and followed for 30 days post infusion.
  ch806:ch806 is a chimeric (part human, part mouse) antibody which recognizes and attaches to a protein called the 806 antigen (a type of EGFR), which is found on the surface of some cancer cells.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 2 | 2 | 2 | 2
hours
  T½α (initial half life) of 111In-ch806 | 10.91 (3.4) | 11.75 (4.4) | 9.34 (8.3) | 8.95 (3.2)
  T½β (terminal half life) of 111In-ch806 | 183.9 (110.2) | 124.5 (9.25) | 125.3 (73.66) | 133.9 (10.79)

6. Secondary Outcome: Mean Volume of the Central Compartment (V1) of 111In-ch806 Following the First Infusion.
Description: as for outcome 5
Time Frame: as for outcome 5
Population: All Patients
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 2 | 2 | 2 | 2
mL | 2963.06 (493.23) | 3060.29 (721.70) | 2902.06 (1064.77) | 4742.42 (169.10)

7. Secondary Outcome: Mean Total Serum Clearance (CL) of 111In-ch806 Following the First Infusion.
Description: as for outcome 5
Time Frame: as for outcome 5
Population: All patients
Measure: Mean (Standard Deviation); unit: mL/hour
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 2 | 2 | 2 | 2
mL/hour | 21.97 (16.59) | 28.58 (8.60) | 30.98 (21.65) | 37.99 (6.47)

8. Secondary Outcome: Mean Area Under the Serum Concentration Curve (AUC) of 111In-ch806 Following the First Infusion.
Description: as for outcome 5
Time Frame: as for outcome 5
Population: All patients
Measure: Mean (Standard Deviation); unit: hour*mg/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 2 | 2 | 2 | 2
hour*mg/mL | 541.17 (371.75) | 566.79 (26.39) | 1438.12 (957.18) | 2269.04 (381.68)

9. Secondary Outcome: Number of Subjects With Best Overall Tumor Response by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Tumor response was evaluated using computed tomography (CT) and categorized according to RECIST at screening (within 4 weeks of study start) and on day 30. Per RECIST, measurable lesions are categorized as follows: Complete Response (CR): complete disappearance of all target lesions; Partial Response (PR): ≥ 30% decrease from baseline in the total measurable tumor burden (TMTB); Progressive Disease (PD): ≥ 20% increase from nadir in TMTB; Stable Disease (SD): not meeting the above criteria.
Time Frame: 30 days
Population: All patients
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 2 | 2 | 2 | 2
Participants
  Stable Disease | 1 | 2 | 1 | 1
  Progressive Disease | 1 | 0 | 1 | 1

10. Secondary Outcome: Number of Patients With Human Anti-chimeric ch806 Antibodies (HACA)
Description: Patients each received a single infusion of 111In-ch806 on Day 0. To assess the secondary endpoint of immune response to ch806, patient serum samples were collected pre-infusion, then weekly until Day 30 (± 2 days) post infusion.
  Human antibody responses against the chimeric antibody (HACA) induced after treatment of patients were analyzed by an enzyme-linked immunosorbent assay (ELISA) technique.
  Patient sera was considered HACA positive if the normalized optical density (OD415) value exceeded a cut-off value of 37.10% (defined as the mean inter-patient baseline normalized OD value +3 SD of pretreatment sera).
Time Frame: 30 days
Population: All patients
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 2 | 2 | 2 | 2
Participants
  HACA positive | 1 | 0 | 0 | 0
  HACA negative | 1 | 2 | 2 | 2

ADVERSE EVENTS:
Time Frame: 30 days
Description: All AEs occurring during the study were documented on the respective case report form (CRF) pages. Events, which occurred after signed informed consent, but before first administration of study drug, were documented on the Pre-existing Signs and Symptom page. Thereafter, they were documented on the Adverse Event page.
  Documentation of AEs includes: date and time of onset and resolution, severity using NCI CTCAE (Version 3.0), frequency, seriousness, related interventions and outcome.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2 | 0/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=2) | Cohort 2 (N=2) | Cohort 3 (N=2) | Cohort 4 (N=2)
increased intracranial pressure (Nervous system disorders) | 1 | 0 | 0 | 0
tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
pain (General disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=2) | Cohort 2 (N=2) | Cohort 3 (N=2) | Cohort 4 (N=2)
anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
syncope (Cardiac disorders) | 0 | 0 | 0 | 1
vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 1
fatigue (General disorders) | 0 | 0 | 1 | 0
lethargy (General disorders) | 0 | 0 | 0 | 1
rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
blood gamma-glutamyl transferase increased (Investigations) | 1 | 0 | 1 | 0
blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 0
hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0
facial paresis (Nervous system disorders) | 1 | 0 | 0 | 0
dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
aphasia (Nervous system disorders) | 0 | 1 | 0 | 0
headache (Nervous system disorders) | 0 | 0 | 0 | 1
insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1
productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
pruritis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No